CLINICAL TRIAL: NCT00104650
Title: A Randomized, Open Label, Active Controlled Study of AMG 162 in Subjects With Advanced Cancer Currently Being Treated With Intravenous Bisphosphonates
Brief Title: Study of AMG 162 in Subjects With Advanced Cancer Currently Being Treated With Intravenous (IV) Bisphosphonates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040114; NCT00121342 (obsolete NCT alias)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Results first posted 2011-01-07 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Bone Metastases in Men With Hormone-Refractory Prostate Cancer; Bone Metastases in Subjects With Advanced Breast Cancer; Bone Metastases in Subjects With Advanced Cancer or Multiple Myeloma
Keywords: Bone Metastases; AMG 162; Bisphosphonates; Solid Tumor Carcinomas; Advanced
MeSH Terms: conditions — Multiple Myeloma | interventions — Denosumab; Amelogenin

ARMS (3):
- IV Bisphosphonates q 4 weeks (Active Comparator): This is an open-label randomization to receive IV bisphosphonate (administered per package insert) every 4 weeks during the treatment phase. If subjects are enrolled into the extension phase, they will receive AMG 162 180mg (SC) every 4 weeks.
  Interventions: Drug: IV Bisphosphonate q 4 weeks
- 180 mg AMG 162 (SC) q 12 weeks (Experimental): This is an open-label randomization to receive 180 mg AMG 162 (SC) every 12 weeks during the treatment phase. If subjects are enrolled into the extension phase, they will continue to receive 180 mg AMG 162 (SC) every 12 weeks.
  Interventions: Genetic: AMG 162 180 mg (SC) q 12 weeks
- 180 mg AMG 162 (SC) q 4 weeks (Experimental): This is an open-label randomization to receive 180 mg AMG 162 (SC) every 4 weeks during the treatment phase. If subject is enrolled into the extension phase, they will continue to receive 180 mg AMG 162 (SC) every 4 weeks.
  Interventions: Genetic: AMG 162- 180 mg q 4 weeks

INTERVENTIONS:
Genetic: AMG 162 180 mg (SC) q 12 weeks — A 180 mg AMG 162 (SC) administered every 12 weeks for 2 doses (Day 1 and wk 13) in the treatment phase. If subjected are enrolled in the extension phase, they will continue to receive a 180 mg AMG 162 (SC) administered every 12 weeks for 9 doses.
  Arms: 180 mg AMG 162 (SC) q 12 weeks
Drug: IV Bisphosphonate q 4 weeks — IV Bisphosphonate (eg pamidronate or zoledronic acid) every 4 weeks for 6 doses as described by package insert during the treatment phase. If enrolled to the extension phase, subject will be assigned to the AMG 162 180mg (SC) every 4 weeks for 26 doses.
  Arms: IV Bisphosphonates q 4 weeks
Genetic: AMG 162- 180 mg q 4 weeks — A 180 mg AMG 162 (SC) administered every 4 weeks for 6 doses in the treatment phase. If subjected are enrolled in the extension phase, they will continue to receive a 180 mg AMG 162 (SC) administered every 4 weeks for 26 doses.
  Arms: 180 mg AMG 162 (SC) q 4 weeks

SUMMARY:
The purpose of this trial is to determine the effectiveness of AMG 162 in reducing urinary N-telopeptide in advanced cancer subjects with bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age with histologically confirmed solid tumor carcinomas (except lung) or multiple myeloma
* Radiographic evidence of 1 or more bone lesions or lytic lesion in myeloma
* Currently receiving IV bisphosphonates
* Urinary N-Telopeptide (uNTx) greater than 50 nM BCE/mM creatinine
* Eastern Cooperative Oncology Group (ECOG) 0, 1 or 2

Exclusion Criteria:

* More than 2 prior skeletal related events (SRE)
* Known brain metastases
* Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw
* Active dental or jaw conditions which requires oral surgery
* Non-healed dental/oral surgery
* Prior administration of AMG 162
* Evidence of impending fracture in weight bearing bones
* Pregnancy or breastfeeding. Subjects must be surgically sterile, postmenopausal, or must agree to use effective contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Fizazi K, Lipton A, Mariette X, Body JJ, Rahim Y, Gralow JR, Gao G, Wu L, Sohn W, Jun S. Randomized phase II trial of denosumab in patients with bone metastases from prostate cancer, breast cancer, or other neoplasms after intravenous bisphosphonates. J Clin Oncol. 2009 Apr 1;27(10):1564-71. doi: 10.1200/JCO.2008.19.2146. Epub 2009 Feb 23. PMID 19237632
- [Result] Fizazi K, Bosserman L, Gao G, Skacel T, Markus R. Denosumab treatment of prostate cancer with bone metastases and increased urine N-telopeptide levels after therapy with intravenous bisphosphonates: results of a randomized phase II trial. J Urol. 2009 Aug;182(2):509-15; discussion 515-6. doi: 10.1016/j.juro.2009.04.023. Epub 2009 Jun 13. PMID 19524963
- [Derived] Jakob T, Tesfamariam YM, Macherey S, Kuhr K, Adams A, Monsef I, Heidenreich A, Skoetz N. Bisphosphonates or RANK-ligand-inhibitors for men with prostate cancer and bone metastases: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 3;12(12):CD013020. doi: 10.1002/14651858.CD013020.pub2. PMID 33270906
- [Derived] Fizazi K, Bosserman L, Gao G, Skacel T, Markus R. Denosumab treatment of prostate cancer with bone metastases and increased urine N-telopeptide levels after therapy with intravenous bisphosphonates: results of a randomized phase II trial. J Urol. 2013 Jan;189(1 Suppl):S51-7; discussion S57-8. doi: 10.1016/j.juro.2012.11.022. PMID 23234632
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 2 December 2004 through 30 March 2007
Groups:
- Bisphosphonate IV Q4W: Open-label intravenous (IV) bisphosphonate once every 4 weeks (Q4W)
- Denosumab 180 mg Q12W: Open-label denosumab 180 mg by subcutaneous injection once every 12 weeks (Q12W)
- Denosumab 180 mg Q4W: Open-label denosumab 180 mg by subcutaneous injection once every 4 weeks (Q4W)
Period: Treatment Period (25 Weeks)
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Started | 37 | 36 | 38
Received Investigational Product | 35 | 35 | 38
Completed | 25 | 25 | 28
Not Completed | 12 | 11 | 10
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Death | 7 | 5 | 6
Not completed — Disease progression | 2 | 3 | 2
Not completed — Ineligibility determined | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0
Period: Follow-up Period
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Started | 25 | 25 | 28
Completed | 14 | 12 | 18
Not Completed | 11 | 13 | 10
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 3
Not completed — Death | 6 | 6 | 4
Not completed — Disease progression | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 180 mg Q4W | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Total
Number analyzed (Participants) | 38 | 37 | 36 | 111
Age Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (10.7) | 61.6 (11.7) | 65.3 (12.7) | 62.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 19 | 56
  Male | 19 | 19 | 17 | 55
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 22 | 22 | 19 | 63
  Black or African American | 0 | 0 | 1 | 1
  Hispanic or Latino | 16 | 13 | 15 | 44
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Other | 0 | 0 | 1 | 1
Cancer Type Stratification Factor [Number; unit: Participants]
  Breast cancer | 16 | 16 | 14 | 46
  Prostate cancer | 17 | 17 | 16 | 50
  Mutiple myeloma | 2 | 3 | 4 | 9
  Other solid tumor | 3 | 1 | 2 | 6
Urinary N-telopeptide (uNTx) Level [Mean (Standard Deviation); unit: nmol/mmol] — Corrected for urine creatinine (uNTx/Creatinine)
  nmol/mmol | 149.94 (147.20) | 149.88 (176.28) | 175.15 (208.87) | 158.01 (177.11)
Serum C-Telopeptide (CTx) [Mean (Standard Deviation); unit: ng/mL] | 1.12 (1.18) | 1.40 (1.93) | 1.34 (1.27) | 1.28 (1.48)

OUTCOME MEASURES:

1. Primary Outcome: uNTx (Corrected by Creatinine) < 50 Nmol/mmol at Week 13
Description: Urinary N-telopeptide (uNTx) corrected by creatinine (uNTx/Cr) < 50 nmol/mmol at week 13.
Time Frame: 13 weeks
Population: All participants who are randomized to the treatment phase, receive at least one dose of treatment phase investigational product, and have treatment phase baseline measurements of uNTx and at least one treatment phase post-baseline measurement of uNTx.
Measure: Number; unit: Participants
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Number analyzed (Participants) | 35 | 33 | 36
Participants | 10 | 21 | 28
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for cancer type stratification factor; Odds Ratio (OR) = 12.28, 95% CI [3.35 to 45.03]
Statistical Analysis 2: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; Adjusted for cancer type stratification factor; Odds Ratio (OR) = 5.33, 95% CI [1.74 to 16.36]
Statistical Analysis 3: Comparison: Denosumab 180 mg Q4W; Test type: Superiority or Other; Percentage of participants = 77.8, 95% CI [60.8 to 89.9]
Statistical Analysis 4: Comparison: Denosumab 180 mg Q12W; Test type: Superiority or Other; Percentage of participants = 63.6, 95% CI [45.1 to 79.6]
Statistical Analysis 5: Comparison: Bisphosphonate IV Q4W; Test type: Superiority or Other; Percentage of participants = 28.6, 95% CI [14.6 to 46.3]

2. Secondary Outcome: uNTx (Corrected by Creatinine) < 50 Nmol/mmol at Week 25
Description: Urinary N-telopeptide (uNTX) corrected by creatinine < 50 nmol/mmol at week 25.
Time Frame: 25 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Number analyzed (Participants) | 35 | 33 | 36
Participants | 13 | 21 | 23
Statistical Analysis 1: Comparison: Denosumab 180 mg Q4W; Test type: Superiority or Other; Percentage of participants = 63.9, 95% CI [46.2 to 79.2]
Statistical Analysis 2: Comparison: Denosumab 180 mg Q12W; Test type: Superiority or Other; Percentage of participants = 63.6, 95% CI [45.1 to 79.6]
Statistical Analysis 3: Comparison: Bisphosphonate IV Q4W; Test type: Superiority or Other; Percentage of participants = 37.1, 95% CI [21.5 to 55.1]

3. Secondary Outcome: Percent Change of uNTx (Corrected by Creatinne) From Baseline to Week 25
Description: Percent change from baseline to week 25 urinary N-telopeptide (uNTX) calculated using ((week 25 value - baseline value) / baseline value ) x 100.
Time Frame: Baseline, week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Number analyzed (Participants) | 23 | 25 | 26
Percent change | -32.91 (65.91) | -69.09 (29.97) | -41.68 (118.32)
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; p = 0.388, ANCOVA; Adjusted for the stratum to which participants were originally assigned by the Interactive Voice Response System (IVRS)

4. Secondary Outcome: Time to Reduction of uNTX (Corrected by Creatinine) to <50nmol/mmol
Description: Kaplan-Meier estimate of the median time from enrollment to the 1st occurrence of uNTx below 50 nmol BCE/mmol (corrected by creatinine) up to week 25. For participants whose uNTx does not go below 50 nM BCE/mM creatinine, the time is censored at time of last evaluation of uNTx by week 25.
Time Frame: Day 1, week 25
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Number analyzed (Participants) | 35 | 33 | 36
Days | 65 [8 to 141] | 9 [4 to 11] | 10 [8 to 11]
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; p < 0.001, Regression, Cox; Stratified by cancer type and screening uNTx level; Hazard Ratio (HR) = 3.79, 95% CI [2.01 to 7.15]
Statistical Analysis 2: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; p < 0.001, Regression, Cox; Stratified by cancer type and screening uNTx level; Hazard Ratio (HR) = 4.32, 95% CI [2.23 to 8.36]

5. Secondary Outcome: Duration of Maintaining uNTX (Corrected by Creatinine) < 50nmol/mmol
Description: Time from the 1st occurrence of uNTx below 50 nmol BCE/mmol (corrected by creatinine) to the 1st occurrence of uNTx above 50 nmol BCE/mmol up to week 25. For participants who remained below 50 nmol BCE/mmol, the time is censored at the time of last evaluation of uNTx up to week 25.
Time Frame: Day 1, week 25
Population: Treatment Phase Primary Analysis Subset. Median was not reached in at least 1 treatment arm. In lieu of the median, the number of subject whose uNTX (corrected by creatinine) less than 50nmol/mmol is presented.
Measure: Number; unit: Participants
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Number analyzed (Participants) | 35 | 33 | 36
Participants | 25 | 32 | 35
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; p = 0.006, Regression, Cox; Adjusted for cancer type stratification factor and screening uNTx level; Hazard Ratio (HR) = 0.274, 95% CI [0.110 to 0.687]
Statistical Analysis 2: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; p = 0.001, Regression, Cox; Adjusted for cancer type stratification factor and screening uNTx level; Hazard Ratio (HR) = 0.199, 95% CI [0.076 to 0.523]

6. Secondary Outcome: Percent Change of Serum CTX From Baseline to Week 25
Description: Percent change from baseline to week 25 in Type I serum C-Telopeptide (CTX), calculated using ((week 25 value - baseline value) / baseline value ) x 100.
Time Frame: Baseline, week 25
Population: All participants who are randomized to the treatment phase, receive at least one dose of treatment phase investigational product, and have treatment phase baseline measurements of uNTx and at least one treatment phase post-baseline measurement of uNTx and had available data.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Number analyzed (Participants) | 23 | 25 | 26
Percent change | -40.68 (38.93) | -76.74 (19.74) | -68.39 (36.15)
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; p = 0.056, ANCOVA; Adjusted for the stratum to which participants were originally assigned by the Interactive Voice Response System (IVRS)

7. Secondary Outcome: Time to First Skeletal Related Event
Description: Time from study day 1 to first Skeletal Related Event (SRE), defined as >1 of the following: pathological bone fracture, spinal cord compression, surgery or radiation therapy to bone (including the use of radioisotopes).
Time Frame: Day 1, week 25
Population: All participants exposed to investigational product during the treatment phase. Median was not reached in at least 1 treatment arm. In lieu of the median, the number of subject who experienced a skeletal related event is presented.
Measure: Number; unit: Participants
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Number analyzed (Participants) | 35 | 35 | 38
Participants | 6 | 4 | 2
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; p = 0.105, Regression, Cox; Hazard Ratio (HR) = 0.162, 95% CI [0.018 to 1.465]
Statistical Analysis 2: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; p = 0.430, Regression, Cox; Hazard Ratio (HR) = 0.573, 95% CI [0.143 to 2.289]

8. Secondary Outcome: Skeletal Related Events
Description: Skeletal Related Event (SRE), defined as >1 of the following: pathological bone fracture, spinal cord compression, surgery or radiation therapy to bone (including the use of radioisotopes).
Time Frame: Day 1, week 25
Population: All participants exposed to investigational product during the treatment phase.
Measure: Number; unit: Participants
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Number analyzed (Participants) | 35 | 35 | 38
Participants | 6 | 4 | 2
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; Odds Ratio (OR) = 0.26, 95% CI [0.05 to 1.44]
Statistical Analysis 2: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; Odds Ratio (OR) = 0.36, 95% CI [0.08 to 1.76]

9. Secondary Outcome: Hypercalcemia
Description: Occurrence of hypercalcemia at grade 3 or 4 according to CTCAE v3 criteria
Time Frame: Day 1, week 25
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Number analyzed (Participants) | 35 | 33 | 36
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 25 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Bisphosphonate IV Q4W | Denosumab 180 mg Q12W | Denosumab 180 mg Q4W
Serious Adverse Events (participants affected / at risk) | 19/35 | 16/35 | 21/38
Other Adverse Events (participants affected / at risk) | 33/35 | 29/35 | 29/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisphosphonate IV Q4W (N=35) | Denosumab 180 mg Q12W (N=35) | Denosumab 180 mg Q4W (N=38)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 4
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 3
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 2 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Death (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 3 | 1
Obstruction (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 2 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vaginal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Areflexia (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Epiduritis (Nervous system disorders) | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Kidney enlargement (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Scar (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Radiotherapy to bone (Surgical and medical procedures) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Neurogenic shock (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bisphosphonate IV Q4W (N=35) | Denosumab 180 mg Q12W (N=35) | Denosumab 180 mg Q4W (N=38)
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Angina pectoris (Cardiac disorders) | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 2
Conjunctivitis (Eye disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 1
Constipation (Gastrointestinal disorders) | 6 | 7 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 5
Gastritis (Gastrointestinal disorders) | 5 | 1 | 1
Nausea (Gastrointestinal disorders) | 7 | 8 | 9
Stomatitis (Gastrointestinal disorders) | 4 | 3 | 3
Vomiting (Gastrointestinal disorders) | 6 | 5 | 2
Asthenia (General disorders) | 7 | 8 | 7
Chills (General disorders) | 3 | 0 | 1
Fatigue (General disorders) | 4 | 3 | 5
Mucosal inflammation (General disorders) | 1 | 0 | 2
Oedema peripheral (General disorders) | 1 | 5 | 6
Pyrexia (General disorders) | 0 | 1 | 5
Bronchitis (Infections and infestations) | 1 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 5
Weight decreased (Investigations) | 0 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 12 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 3
Paraesthesia (Nervous system disorders) | 3 | 4 | 6
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 5 | 3 | 1
Insomnia (Psychiatric disorders) | 4 | 1 | 2
Haematuria (Renal and urinary disorders) | 1 | 2 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2
Gynaecomastia (Reproductive system and breast disorders) | 2 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Radiotherapy to bone (Surgical and medical procedures) | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.